CLINICAL TRIAL: NCT06084546
Title: Evaluation of the Adhesive Strength of an Improved Skin Adhesive Hydrogel Formulation Designated KM40C Incorporated in the Geko™ X-W3 Neuromuscular Electrical Stimulator (NMES) Device in Patients With Lower Limb Ulcers
Brief Title: Geko™ KM40C Hydrogel Skin Adhesion Trial (XW-3)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FSK-R&D-002
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Leg Ulcer
Keywords: geko; NMES
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care with geko™ W3 device (No Intervention): Current geko™ device incorporating hydrogel adhesive designated KM40A
- Standard care with geko™ X-W3 (Active Comparator): Next generation geko™ device incorporating new hydrogel adhesive designated KM40C
  Interventions: Device: geko™ X-W3

INTERVENTIONS:
Device: geko™ X-W3 — The geko™ X-W3 is a next generation self adhesive medical device incorporating a new formulation skin adhesive. It is about the size of a wrist watch which attaches to the side of the knee and when switched on, gentle painless electrical pulses are produced which contract the calf muscles and increase blood flow to the lower leg. The only difference between the currently used geko™ W3 device and the new geko™ XW-3 device is the adhesive used to attach each device to the skin.
  Arms: Standard care with geko™ X-W3

SUMMARY:
Hydrogel KM40C is an electrically conductive skin adhesive incorporated in the self-adhesive, geko™ XW-3 neuromuscular electrical stimulation (NMES) device. KM40C has been formulated to adhere to the skin giving good electrical contact for the electrodes, be easy to remove without damaging the skin and be non-irritant. KM40C has been tested for safety in humans, however the skin adhesive performance of this improved hydrogel formulation has not been tested on patients receiving geko™ NMES treatment as an adjunct to standard care for wound management.

The objective of this trial is to evaluate the skin adhesive performance of hydrogel KM40C during clinical use of the geko™ XW-3 NMES device to determine whether skin adhesion is at least equivalent if not superior to the adhesive hydrogel KM40A incorporated in the self-adhesive geko™ W3 device which is currently in use clinically. Both devices are indicated for use to promote wound healing, the geko™ W3 NMES device is UKCA and CE marked whereas the geko™ X-W3 is UK CA marked only.

ELIGIBILITY:
Inclusion Criteria:

1. Adult over 18.
2. Patients who have a lower limb ulcer following evaluation by a Tissue Viability Nurse Specialist
3. Intact healthy skin at the site of geko™ device application.
4. Willing and able to give written informed consent
5. Identified to receive geko™ treatment as an adjunct to standard care for wound management.

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Use of any other neuro-modulation device.
3. Use of a cardiac pacemaker
4. Current use of TENS in the pelvic region, back or legs
5. Contraindication to geko ™ NMES treatment
6. No response to geko ™ NMES i.e. no involuntary rhythmic upward and outward movement of the foot (dorsiflexion) at the maximum tolerable device setting.
7. Participation in any other clinical trial that may interfere with the outcome of either trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Skin Adhesive Strength of Hydrogel KM40C Compared to That of Hydrogel KM40A | 28 days
  Self reported - how well did the geko™ device stick to the patients leg? Scale 1-5, Lowest score indicates best adhesion.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 28 days
  Reporting of the incidence of adverse events , incidence of serious adverse events, incidence of study treatment related adverse events, and the incidence of device related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Collarte, Principal Investigator — St Charles Centre for Health & Wellbeing
Locations (2):
- United Kingdom (2):
  - Central London Community Health Care NHS Trust, London
  - Norfolk Community Health and Care NHS Trust, Norwich

IPD SHARING:
Plan to Share IPD: No